CLINICAL TRIAL: NCT04318067
Title: Melatonin - Production and Release in Children and Adolescents With ADHD and Chronic Sleep Problems and Effects of Melatonin on Sleep
Brief Title: Melatonin in ADHD and Sleep Problems
Acronym: MELAS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Allan Hvolby (Other)
Collaborators: Sygehus Lillebaelt (Other)
Responsible Party: Sponsor-Investigator, Allan Hvolby, Principal Investigator, MD, Ph.D, Region of Southern Denmark
Organization: Region of Southern Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18081070
Record Dates: First submitted 2020-02-14; First posted 2020-03-23 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Attention Deficit Hyperactivity Disorder; Sleep Disorder
Keywords: Melatonin; Attention Deficit Hyperactivity Disorder; Sleep problems; Dim Light Melatonin Onset
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Sleep Wake Disorders; Parasomnias | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sleep problems i Attention Deficit Hyperactivity Disorder (Experimental): Children age 6 to 12 years having ADHD and Sleeping problem will be treated with Melatonin 3 mg one a day (before bedtime)
  Interventions: Drug: Melatonin 3 mg

INTERVENTIONS:
Drug: Melatonin 3 mg — Melatonin 3 mg is given ones a day - at bedtimes for 6 month

SUMMARY:
Treatment with melatonin is often initiated on an insufficient basis as it has not been established prior to starting the treatment whether or not the child had delayed release of endogenous melatonin. At the clinic, it has furthermore been observed that the length of time a child experiences an effect of melatonin treatment varies substantially.

In a clinical context, treatment with melatonin is used increasingly (www.Medstat.dk). However, there is no tradition in Denmark for measuring the endogenous melatonin level before initiating such treatment. Hence there is no way of knowing to what extent the sleep problems were indeed caused by delayed melatonin release.

There seem to be no studies on the difference in the effect of melatonin treatment of children and adolescents depending on whether or not they have delayed DLMO. Likewise, there are no studies including adolescents.

As can be seen, it is important to gain more knowledge about the normal release of melatonin, and the release of melatonin in a group of children and adolescents with a variety of psychiatric diagnoses. It is also essential to investigate whether there are any differences in the release of melatonin in children and adolescents with chronic sleep onset problem and children and adolescents who do not have sleep problems.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-13 years referred to the child and adolescent psychiatric department for examination/treatment for ADHD
* Verified Cronical Sleep Problems
* Measured Dim Light Melatonin Onset

Exclusion Criteria:

* IQ below 70
* Autism Disorder
* Actual or former treated with Melatonin
* Allergy to melatonin

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Sleep onset Latency (SOL) | 6 month
  How long time does the child use falling asleep after lights out
Sleep onset | 6 month
  Time where child falls asleep
Total Sleep time | 6 month

SECONDARY OUTCOMES:
Attention Deficit Hyperactivity Disorder - Scale Score (ADHD-RS) | 6 month
  A Scale Score measuring ADHD symptoms on a 4 point Likert Scale (0-3) . 18 Question with a Total max score of 54, Total minimum Score is 0 . Higher score is more symptoms.
Weiss Functional Impairment Rating Scale (WFIRS) | 6 month
  Evaluation on different Quality of Life (QoL) scores. 50 Question Measuring QoL in School, Family setting and Social activities on a 4 Point Likert Scale (0-3) with af total max score om 150 (minimum 0) - A higher score is more difficulties and lower Quality of Life
Dundee Difficult Times of the Day Scale (D-DTODS) | 6 month
  On a 4 point Likert scale (1-4) the instrument asses the impact on Child and Family Self-Esteem and Quality of Life . Total max is 40 points and indicates low QoL and Minimum score is 10 and indicate Normal functioning and High QoL
Side effect Rating Scale | 6 month
  Registration of 17 known possible Side Effekts on a Likert Scale 0-9 point each, With a total score of 153 points which indicate many and serious Side effect and a minimum of 0 , which indicate Zero side effects

CONTACTS AND LOCATIONS:
Overall Officials: Allan Hvolby, MD, Ph.D, Principal Investigator — Child and adolescent Psychiatric department, South Jutland
Locations (1):
- Child and Adolescent Psychiatric department, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: No